CLINICAL TRIAL: NCT07400237
Title: Laparoscopic Ultrasound Versus Fluorescence Cholangiography in Technically Challenging Laparoscopic Cholecystectomy. Multicenter Comparative Study
Brief Title: Laparoscopic Ultrasound Versus Fluorescence Cholangiography in Technically Challenging Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari Integral (Other)
Collaborators: Hospital Moisés Broggi de Sant Joan Despí, Barcelona (Unknown); Hospital Clínico Universitario de Valencia (Other); Hospital Germans Tríes i Pujol de Badalona (Unknown); Hospital Joan XXIII, Tarragona (Unknown); Consorcio Parc de Salut Mar, Hospital del Mar (Unknown); Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24/49
Record Dates: First submitted 2026-01-16; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Cholecystectomy
Keywords: laparoscopic cholecystectomy; laparoscopic ultrasound; fluorescence cholangiography; indocyanine green; biliary injury prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complex laparoscopic cholecystectomy (Other): Laparoscopic cholecystectomy with anticipated technical difficulty
  Interventions: Diagnostic Test: Laparoscopic ultrasound (LUS) and fluorescence cholangiography with indocyanine green (ICG)

INTERVENTIONS:
Diagnostic Test: Laparoscopic ultrasound (LUS) and fluorescence cholangiography with indocyanine green (ICG) — Two intraoperative imaging modalities will be applied: laparoscopic ultrasound (LUS) and fluorescence cholangiography with indocyanine green (ICG), for the identification of biliary anatomy in technically challenging laparoscopic cholecystectomy. All enrolled subjects will undergo both LUS and ICG during the index procedure, following a standardized sequence, in order to allow intra-subject comparison. LUS will be performed first, followed by fluorescence cholangiography prior to Calot's triangle dissection.

SUMMARY:
This is a multicenter, prospective, interventional clinical trial designed to evaluate and compare two intraoperative imaging modalities: laparoscopic ultrasound (LUS) and fluorescence cholangiography with indocyanine green (ICG), for the identification of biliary anatomy in technically challenging laparoscopic cholecystectomy. All enrolled subjects will undergo both LUS and ICG during the index procedure, following a standardized sequence, in order to allow intra-subject comparison. LUS will be performed first, followed by fluorescence cholangiography prior to Calot's triangle dissection.

The primary endpoint is the successful identification of the critical junction. Secondary endpoints include visualization of individual biliary structures, time to visualization, total operative time, intraoperative and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Written informed consent provided.
3. Indication for laparoscopic cholecystectomy with anticipated technical difficulty due to one or more of the following:

   * Acute cholecystitis.
   * Previous cholangitis, pancreatitis, or endoscopic retrograde cholangiopancreatography.
   * Prior upper abdominal surgery.
   * Obesity (Body Mass Index ≥ 30 kg/m²).

Exclusion Criteria:

1. Known allergy to ICG or iodine.
2. Pregnancy or breastfeeding.
3. High risk of choledocholithiasis (ESGE guidelines).
4. Thyroid disease.
5. Suspected gallbladder malignancy.
6. ASA class IV-V.
7. Chronic kidney disease stage > IIIb.
8. Planned open cholecystectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clear intraoperative identification of the junction between the cystic duct, the common hepatic duct, and the common bile duct | Intraoperative
  This intraoperative visualization will be assessed separately for laparoscopic ultrasound (LUS) and indocyanine green fluorescence cholangiography (ICG) and recorded as a binary outcome (yes/no) for each technique in each patient using a standardized intraoperative assessment form completed by the operating surgeon.
  Laparoscopic ultrasound will be performed first, followed by indocyanine green fluorescence cholangiography, according to a predefined and standardized intraoperative sequence.
  Intraoperative photographic documentation will be obtained for each imaging modality to objectively demonstrate the visualization of the critical biliary junction.
  Results will be reported as the proportion of patients with successful visualization for each modality and compared using an intra-subject analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Complex Hospitalari Universitari Moisès Broggi, Consorci Sanitari Integral, Sant Joan Despí, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No